CLINICAL TRIAL: NCT01688427
Title: Perinatal Nurse Home Visiting Enhanced With mHealth Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NA_00051481; 1R01HD071771-01 (NIH)
Record Dates: First submitted 2012-09-10; First posted 2012-09-19 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Domestic Violence; Intimate Partner Violence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard IPV Assessment (Experimental): Test the effectiveness of the eMOCHA DOVE application using mHealth technology for routine assessment of IPV vs. Pencil and paper.
  Interventions: Behavioral: Standard IPV Assessment
- Standard DOVE intervention (Experimental): The standard DOVE intervention has already been developed and tested (NR009093). The standard DOVE intervention is a brochure based 10 minute intervention that the home visitor reviews with the women. It consists of information about IPV, its effects on pregnancy and infant health, community resources and a plan for individual safety options. For the eMOCHA DOVE intervention, the DOVE 10 minute brochure intervention will be converted from the paper format to a visually colorful interactive presentation loaded into the home visitor device using the eMOCHA application. The format will be completely activated and implemented by the women. She uses small ear buds and a touch screen, so how she responds and interacts with the media enhanced eMOCHA DOVE intervention is private.
  Interventions: Behavioral: Standard IPV Assessment; Behavioral: Standard DOVE Intervention

INTERVENTIONS:
Behavioral: Standard IPV Assessment — Test the effectiveness of the eMOCHA DOVE application using mHealth technology for routine assessment of IPV vs. Pencil and paper at enrollment, delivery, and 2 months post birth.
Behavioral: Standard DOVE Intervention — Intervention will be administered via eMOCHA tablet vs. home visitor over 6 sessions in 6 months.
  Arms: Standard DOVE intervention

SUMMARY:
This research is being done to test whether mobile technology will reduce possible communication barriers between women and their home visitor; to improve assessing for health problems that could affect their pregnancy; to help in the delivery of information and actions to improve the health of the woman and their child.

DETAILED DESCRIPTION:
This study addresses PA-11-104 calling for Reducing Health Disparities among Minority and Underserved Children. The Institute of Medicine, World Health Organization and Centers for Disease Control and Prevention recognize that prenatal home visitation, which improves the well-being of mother and children, presents an opportunity to provide early intervention to reduce intimate partner violence (IPV) and the impact the exposure has on the children. Major challenges for nurses and other home visitors (HV) are to accurately identify abused women and facilitate their accessing resources needed to change their situation. HVs often find it difficult to assess and intervene for IPV in the intimacy of home settings. The use of mHealth technology may increase the sensitivity of screening instruments and reduce communication barriers between HVs and clients regarding IPV, as well as enhance implementation of IPV interventions and allow for a more standard delivery of an intervention. Building on the successful trial testing the DOVE IPV intervention in prenatal home visiting programs (NR009093), the investigators propose to test mHealth technology using an open-source application, eMOCHA, to improve assessment of IPV and to deliver the DOVE intervention. The proposed eMOCHA DOVE study will first (Specific Aim/Phase 1) compare sensitivity and specificity of two different approaches for IPV assessment; paper and pencil versus the eMOCHA mHealth technology. Phase 2 (Aim 2) will compare effectiveness of the DOVE intervention delivered in standard form (paper brochure) versus mHealth eMOCHA DOVE application. In Phase 1 women enrolled in a perinatal home visiting program and consenting to the study, will be randomized to one of the two assessment groups and assessed for IPV at enrollment, birth and 2 months post birth. Women who are IPV positive (IPV+) at any of the assessment times will be re-randomized to receive the DOVE intervention by one of the two approaches. 1600 Medicaid eligible pregnant women in a perinatal home visiting program (800 from urban Baltimore and 800 from rural Virginia) will be recruited for Phase I and 400 IPV+ women (200 from each site) for Phase II. Women participating in Phase 2 will receive 6 home visit interventions over 6 months. Maternal outcomes related to IPV and mental health and selected infant outcomes will be collected at enrollment, 3, 6, 12, and 18 months after entry into Phase 2. Specific Aim 1 will use logistic and linear regression models to examine the proportion of women experiencing IPV through mHealth technology versus paper and pencil on the same validated assessments. Specific Aim 2 (comparing effectiveness of two intervention administrations) will be assessed with logistic and linear regression models for categorical (proportion abused and premature infants) and continuous outcome variables (e.g. depression, frequency and severity of physical, psychological, sexual IPV, use of community resources) respectively. Study findings will assist nurse home visitation programs to use best approaches for routine assessment of IPV and implement empowerment interventions to reduce IPV and improve maternal infant health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women in Baltimore, Virginia, and Missouri if needed.
* Speak English or Spanish
* Eligible for home visitation.

Exclusion Criteria:

* Women who begin participation in a perinatal home visiting program after the baby is born.
* Women who do not speak English or Spanish.

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 433 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Change in IPV assessments | Screening and at 2 months post-birth.
  Instances of intimate partner violence (IPV).

SECONDARY OUTCOMES:
Change in use of safety behaviors | Baseline and end of study (approximately 18 months post-birth)
  Record the number of pregnant/parenting women using safety behaviors (including mental health and other community resources).
Change in number of safety behaviors | Baseline and end of study (approximately 18 months post-birth)
  Record the aggregate number of services (including mental health and other community resources).

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis W Sharps, PhD, Principal Investigator — Johns Hopkins University, School of Nursing; Linda Bullock, PhD, RN, Principal Investigator — University of Virginia
Locations (1):
- Johns Hopkins University, School of Nursing, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Bacchus LJ, Bullock L, Sharps P, Burnett C, Schminkey DL, Buller AM, Campbell J. Infusing Technology Into Perinatal Home Visitation in the United States for Women Experiencing Intimate Partner Violence: Exploring the Interpretive Flexibility of an mHealth Intervention. J Med Internet Res. 2016 Nov 17;18(11):e302. doi: 10.2196/jmir.6251. PMID 27856405